CLINICAL TRIAL: NCT06201247
Title: Safety and Efficacy of Universal Off-the-shelf CAR-NK Cells Targeted CD123 (JD123 Injection) in the Treatment of Refractory or Relapsed CD123-positive Acute Myeloid Leukemia
Brief Title: Off-the-shelf CD123 CAR-NK for R/R AML
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Xiao-Jun Huang, Professor, Peking University People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023PHD016-001
Record Dates: First submitted 2023-12-30; First posted 2024-01-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Acute Myeloid Leukemia, in Relapse; Acute Myeloid Leukemia Refractory
Keywords: Acute Myeloid Leukemia; CAR-NK
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Intervention Model Description: 3+3 Phase I
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: Experimental: JD123 injection. (Experimental): The relapsed/refractory AML patients will receive JD123 injections up to 3 dose levels (5.0×108 cells/dose，1.5×109 cells/dose，3.0×109 cells/dose) after FC chemotherapy.
  Interventions: Drug: JD123 injection

INTERVENTIONS:
Drug: JD123 injection — JD123 injection is an universal Off-the-shelf CD123-targeted chimeric antigen receptor modified natural killer cells (CAR-NK) therapy derived from a healthy donor.

SUMMARY:
This is a single-centre, single-arm, open-label, first-in-human (FIH) study to evaluate the safety, tolerability and preliminary efficacy of universal Off-the-shelf CAR-NK cells targeted CD123 (JD123 injection) in the treatment of refractory or relapsed CD123-positive acute myeloid leukemia (AML).

DETAILED DESCRIPTION:
This is a dose-escalation study of CD123-targeted chimeric antigen receptor modified natural killer cells (CAR-NK) derived from a healthy donor. The relapsed/refractory AML patients will receive FC (F, Fludarabine, C, Cyclophosphamide) chemotherapy followed by infusion of JD123 injections. No graft-versus-host disease (GVHD) prevention will be conducted before or after infusion. Dose-limiting toxicity, incidence of adverse events, disease response and PK/PD will be detected post-infusion.

ELIGIBILITY:
Inclusion criteria:

1. Age ≥ 18 years old, no gender or race;
2. Expected survival period ≥ 3 months;
3. Eastern Cooperative Oncology Group (ECOG) performance status score of 0 to 2;
4. The diagnosis of AML with bone marrow biopsy, immunohistochemistry or Flow cytometry definitively positive for CD123 and met the following criteria:

   A. Diagnostic criteria for relapsed AML: after complete remission (CR), leukemia cells reappeared in peripheral blood or blast cells in bone marrow ≥ 5% (except for other reasons such as bone marrow regeneration after consolidation chemotherapy) or extramedullary leukemia cell infiltration; B. Diagnostic criteria for refractory AML: naive patients who were ineffective after 2 courses of standard regimens; patients relapsed within 12 months who underwent consolidation and intensive therapy after CR; patients relapsed after 12 months but were ineffective after conventional chemotherapy; Patients with two or more relapses; patients with persistent extramedullary leukemia; Patients relapsed after allogeneic hematopoietic stem cell transplantation (allo-HSCT) C. Minimal Residual Disease (MRD) positive only or relapse: Patient is minimal residual disease (MRD) positive, as assessed on bone marrow aspirate (BMA) by Multiparameter Flow Cytometry (MFC) at time of Treatment Eligibility assessment.
5. Adequate organ function:

A. Liver function: ALT≤3×ULN, AST≤3×ULN, total bilirubin≤2×ULN; B. Coagulation function: international normalized ratio (INR) or activated partial thromboplastin time (APTT) ≤ 1.5×ULN; C. Renal function: serum creatinine≤1.5×ULN or creatinine clearance rate ≥30mL/min; D. Cardiac function: Left ventricular ejection fraction (LVEF) ≥ 50%; 6. Women of child-bearing potential and all male participants must use effective methods of contraception for at least 12 months after infusion.; 7. Informed Consent/Assent: All subjects must have the ability to understand and the willingness to sign a written informed consent.

Exclusion Criteria:

1. Active Central nervous system leukemia;
2. Known contraindication to the protocol defined lymphodepleting chemotherapy regimen of fludarabine/cyclophosphamide;
3. Systemic use of hormones within 4 weeks prior to enrollment (except for patients with inhaled corticosteroids);
4. Any active infection requiring systemic therapy by intravenous infusion within 14 days prior to the first dose of study drug, including: HBV, HCV, HIV, syphilis infection, or active pulmonary tuberculosis.
5. History of hypersensitivity reactions to murine protein-containing products, or macromolecular biopharmaceuticals such as antibodies or cytokines;
6. Patients cannot guarantee effective contraception (condom or contraceptives, etc.) within 1 years after enrollment;
7. Women who are pregnant (urine/blood pregnancy test positive) or lactating;
8. Suffering from a serious autoimmune disease or immunodeficiency disease; 9 Suffering from mental illness;

10. Known alcohol dependence or drug dependence; 11. According to the investigator's judgment, the patient has other unsuitable grouping conditions.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2023-12-30 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
1-month DLTs | 1-month
  Dose limiting toxicities (DLTs)

SECONDARY OUTCOMES:
3-month CR/CRi | 3-month
  Complete response (CR) or Complete remission with incomplete recovery(CRi)
1-year PFS | 1-year
  Progression free survival(PFS)
1-year OS | 1-year
  Overall Survival (OS)
1-year MRD(-) | 1-year
  Proportion of subjects with minimal-residual disease (MRD) negative response
3-month AUC | 3-month
  The area under the concentration time-curve (AUC) of CD123-CAR-NK cells
3-month Peak | 3-month
  Peak levels of CD123-CAR-NK cells (maximum concentration or Cmax)

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China